CLINICAL TRIAL: NCT02904720
Title: Prevalence and Consequences of Vitamin D Deficiency in Pregnant Women in Switzerland
Acronym: PCVDDPWS
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Significantis GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2015-00063
Record Dates: First submitted 2016-09-08; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Pregnancy
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the prevalence of vitamin D deficiency among the population of pregnant women receiving prenatal care and giving birth at the investigators' clinic. The further purposes are to identify the population at risk for vitamin D deficiency and to analyse whether vitamin D deficiency is associated with pregnancy complications.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending prenatal care at our clinic who had a vitamin D blood-testing at admission

Exclusion Criteria:

* Pregnant women lost to follow-up, Birth outside our clinic

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the pregnant women attending prenatal care and giving birth at birth at our clinic
Sampling Method: Non-Probability Sample
Enrollment: 1199 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of vitamin D deficiency | Between the 1th and the 36th week of pregnancy
  Number of patients with vitamin D deficiency after testing of vitamin D blood level at admission for prenatal care in our clinic

SECONDARY OUTCOMES:
BMI as a risk factor for vitamin D deficiency | Between the 1th and the 36th week of pregnancy
  Presence of an association between the patient's BMI and their vitamin D blood level?
Ethnicity as a risk factor for vitamin D deficiency | Between the 1th and the 36th week of pregnancy
  Presence of an association between the patient's ethnicity and their vitamin D blood level?
Age as risk factor for vitamin D deficiency | Between the 1th and the 36th week of pregnancy
  Presence of an association between the patient's age and their vitamin D blood level ?
Period of the year as risk factor for vitamin D deficiency | Between the 1th and the 36th week of pregnancy
  Presence of an association between the period of the year at the time of the blood testing and the vitamin D blood level?
Smoking Status as risk factor for vitamin D deficiency | Between the 1th and the 36th week of pregnancy
  Presence of an association between the patient's smoking status and the vitamin D blood level ?
Association between vitamin D blood level and gestational diabetes mellitus | Between the 1th and the 36th week of pregnancy
  Presence of an association between the vitamin D blood level and the occurrence of gestational diabetes mellitus?
Association between vitamin D blood level and gestational hypertension and preeclampsia | Between the 1th and the 36th week of pregnancy
  Presence of an association between the vitamin D blood level and the occurrence of gestational hypertension and preeclampsia ?

OTHER OUTCOMES:
Association between vitamin D blood level and the mode of delivery at birth | At delivery time
  Presence of an association between the vitamin D blood level and the mode of delivery (Vaginal delivery, instrumentalized delivery, primary and secondary cesarean)?
Association between vitamin D blood level and the gestational age at delivery | At delivery time
  Presence of an association between the vitamin D blood level and the gestational age at delivery? Occurrence of preterm birth (before 37W) or postterm birth (after 40W)?
Association between vitamin D blood level and newborn growth | From week 1 until birth
  Presence of an association between vitamin D blood level and the occurrence of intrauterin growth retardation or small-for-gestational age child? With assessment of measure like length, weight, head perimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Surbek, Professor, Study Director — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christoph P, Challande P, Raio L, Surbek D. High prevalence of severe vitamin D deficiency during the first trimester in pregnant women in Switzerland and its potential contributions to adverse outcomes in the pregnancy. Swiss Med Wkly. 2020 May 28;150:w20238. doi: 10.4414/smw.2020.20238. eCollection 2020 May 18. PMID 32502277